CLINICAL TRIAL: NCT06230055
Title: Clinical Outcome and Quality of Life of Intrathecal Chemotherapy Through Ommaya Reservoir in Combination With Systematic Chemotherapy Versus Systematic Chemotherapy Upon Her-2 Negative Breast Cancer With Leptomeningeal Metastasis (CONQUER)
Brief Title: Intrathecal Chemotherapy Through Ommaya Reservoir Upon Her-2 Negative Breast Cancer With Leptomeningeal Metastasis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, Chief physician, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONQUER
Record Dates: First submitted 2023-12-29; First posted 2024-01-29 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: HER2-negative Breast Cancer; Leptomeningeal Metastasis
MeSH Terms: conditions — Meningeal Carcinomatosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intrathecal chemotherapy through Ommaya reservoir in combination with systematic chemotherapy (Experimental): Intrathecal chemotherapy through Ommaya reservoir: including MTX(10-12mg, q1-3w), thiotepa(10mg, q1-3w), cytarabine(30mg/m2, q1-3w), cytarabine liposome(50mg, q1-3w), pemetrexed(50mg, q1-3w), or DS8201(The frequency and cycle of drug administration are determined based on the results of the Phase I/II clinical trial of intrathecal injection of DS8201 in our center).
  Systematic chemotherapy: including capecitabine(1000mg/m2 bid, d1-14, q3w, po), gemcitabine(1000mg/m2, d1,8, q3w, ivgtt), vinorelbine(60mg/m2, qw, po), docetaxel(75mg/m2, d1, q3w, ivgtt),Nab-paclitaxel(125mg/m2, d1,8, q3w, ivgtt), iribrin(1.4mg/m2, d1,8, q3w, ivgtt), DS8201(5.4mg/kg, d1, q3w, ivgtt), sacituzumab govitecan(10mg/kg, d1,8, q3w, ivgtt) or SKB264(5mg/kg, d1, q2w, ivgtt).
  Interventions: Device: Ommaya reservoir; Drug: Systematic chemotherapy; Drug: Intrathecal chemotherapy
- systematic chemotherapy (Active Comparator): Systematic chemotherapy: including capecitabine(1000mg/m2 bid, d1-14, q3w, po), gemcitabine(1000mg/m2, d1,8, q3w, ivgtt), vinorelbine(60mg/m2, qw, po), docetaxel(75mg/m2, d1, q3w, ivgtt),Nab-paclitaxel(125mg/m2, d1,8, q3w, ivgtt), iribrin(1.4mg/m2, d1,8, q3w, ivgtt), DS8201(5.4mg/kg, d1, q3w, ivgtt), sacituzumab govitecan(10mg/kg, d1,8, q3w, ivgtt) or SKB264(5mg/kg, d1, q2w, ivgtt).
  Interventions: Drug: Systematic chemotherapy

INTERVENTIONS:
Device: Ommaya reservoir — Intrathecal chemotherapy through Ommaya reservoir
  Arms: intrathecal chemotherapy through Ommaya reservoir in combination with systematic chemotherapy
Drug: Systematic chemotherapy — Systematic chemotherapy: including capecitabine(1000mg/m2 bid, d1-14, q3w, po), gemcitabine(1000mg/m2, d1,8, q3w, ivgtt), vinorelbine(60mg/m2, qw, po), docetaxel(75mg/m2, d1, q3w, ivgtt),Nab-paclitaxel(125mg/m2, d1,8, q3w, ivgtt), iribrin(1.4mg/m2, d1,8, q3w, ivgtt), DS8201(5.4mg/kg, d1, q3w, ivgtt), sacituzumab govitecan(10mg/kg, d1,8, q3w, ivgtt) or SKB264(5mg/kg, d1, q2w, ivgtt).
Drug: Intrathecal chemotherapy — Intrathecal chemotherapy through Ommaya reservoir: including MTX(10-12mg, q1-3w), thiotepa(10mg, q1-3w), cytarabine(30mg/m2, q1-3w), cytarabine liposome(50mg, q1-3w), pemetrexed(50mg, q1-3w), or DS8201(The frequency and cycle of drug administration are determined based on the results of the Phase I/II clinical trial of intrathecal injection of DS8201 in our center).
  Arms: intrathecal chemotherapy through Ommaya reservoir in combination with systematic chemotherapy

SUMMARY:
This is a prospective, multicenter, randomized controlled, open-label investigator-initiated clinical study to evaluate the clinical efficacy and quality of life of intrathecal chemotherapy through Ommaya reservoir in combination with systematic chemotherapy versus systemic chemotherapy alone in patients with Her-2 negative breast cancer with leptomeningeal metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years or above;
2. Can understand the purpose of clinical trials and the benefits and risks, voluntarily participate in and sign the informed consent
3. The physical status score of the Eastern Oncology Consortium (ECOG) was ≤3;
4. HER2-metastatic breast cancer confirmed histologically or cytologically (HER2- is defined as either a standard immunohistochemical (IHC) test result of 0 or 1+, or an IHC test result of 2+ and a negative ISH test result);
5. Failure of standard treatment, or intolerance to standard treatment;
6. pial metastasis is present, which is defined as meningeal metastasis confirmed by malignant tumor cells found in cerebrospinal fluid cytology; Or clinical symptoms/signs suggest meningeal metastasis, and brain MRI suggests pia enhancement;
7. The function of major organs was good, which was confirmed by the following laboratory tests during the screening period:

   Platelet count ≥80*10^9/L

   Hemoglobin ≥8g/L

   Neutrophil count ≥1.5*10^9/L

   Serum creatinine ≤1.5*ULN

   ALT and AST≤ 3*ULN (if liver metastases are present, ALT and AST≤5*ULN)

   Serum total bilirubin ≤1.5*ULN

   International Standardized ratio (INR) and Activated partial thromboplastin time (APTT) ≤1.5*ULN
8. NYHA cardiac function grade ≤II, no obvious abnormality in ECG, or no clinical significance according to the investigators;
9. Voluntary compliance with the trial protocol during the study period and regular follow-up;
10. For all women of childbearing age, fertile men or their spouses who did not plan to have children or donate sperm during the entire trial period until 6 months after the last dose, or who voluntarily took effective contraception, the blood/urine pregnancy test results of female patients of childbearing age within 7 days before enrollment were negative.
11. Subjects who have recovered from non-hematological toxicity from the last treatment (CTCAE≤ class 1, except for special conditions such as "alopecia") before first administration, and who the investigator determines that the corresponding AE does not pose a safety risk.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Patients with acute and chronic infections, or with other serious diseases at the same time, were judged not suitable for this study;
3. Other malignant tumors within 5 years (except the following cases: cured skin basal cell carcinoma, cervical carcinoma in situ, thyroid papillary carcinoma; A second primary cancer that has been eradicated and has not recurred within five years; Both primary cancers are expected to benefit from this study. Investigators have identified the primary tumor source of the metastases);
4. Mental illness or mental disorder, poor compliance can not cooperate with and describe treatment response;
5. There are serious organic diseases or major organ failure, such as decompensated heart and lung failure, which can not tolerate treatment;
6. Patients with bleeding tendency;
7. Patients who have received organ transplants;
8. Patients taking adrenal corticosteroids or immunosuppressants for a long time;
9. Intracranial hemorrhage unrelated to tumor disease;
10. Patients with central nervous system complications requiring urgent treatment;
11. Test group: subjects who could not collect CSF;
12. The subject has a history of immunodeficiency, including HIV testing positive, or other acquired or congenital immunodeficiency diseases;
13. Active viral hepatitis B (HBsAg positive with HBV DNA≥500 IU/mL) or hepatitis C. Among hepatitis C antibody positive subjects, only those whose polymerase chain reaction showed negative HCV RNA were eligible for enrollment (chronic hepatitis B or chronic hepatitis C patients with stable disease receiving standard antiviral therapy were eligible for enrollment);
14. The subject has a serious cardiovascular clinical disease or symptom, including:

    Congestive heart failure

    History of unstable angina;

    myocardial infarction within the past six months;

    Clinically significant malignant arrhythmias (except atrial fibrillation and paroxysmal supraventricular tachycardia);

    Subjects had clinically significant prolonged QTcF

    High blood pressure that is not well controlled;
15. The researcher believes that the patient has other conditions that are not suitable for participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Neural progression-free survival (NPFS) | Six months after the last patient was enrolled
  Clinical outcome of intrathecal chemotherapy through Ommaya reservoir in combination with systematic chemotherapy versus systematic chemotherapy Upon Her-2 negative breast cancer with leptomeningeal metastasis: Neural progression-free survival (NPFS) calculated from the randomized date until first observation of meningeal metastasis progression (LM-PD) or death (whichever occurs earlier). Neural progression, according to the RANO-LM criteria, is defined as: neurological examination/worsening of symptoms, or CSF cytological progression, or imaging progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center; Department of Oncology, Shanghai Medical College, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No